CLINICAL TRIAL: NCT00522522
Title: Naturalistic Study to Evaluate the Utilization of Care Services Associated to the Diagnostic Process of Any Kind of Epilepsy Until Being Confirmed (EPILIVE Study)
Brief Title: Naturalistic Study to Evaluate the Utilization of Care Services Associated to the Diagnostic Process of Any Kind of Epilepsy
Status: Completed | Type: Observational
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: N01292; EPILIVE
Record Dates: First submitted 2007-08-27; First posted 2007-08-29 (Estimated); Last update posted 2012-05-30 (Estimated); Status verified 2012-05

CONDITIONS: Epilepsy
Keywords: Naturalistic, retrospective, utilization of care services, diagnosis, epilepsy
MeSH Terms: conditions — Epilepsy; Disease

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Naturalistic, multicentre, epidemiological study to evaluate the care services used during the process of diagnosis of any kind of epilepsy. Data about services since first seizure until confirmed diagnosis will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes 16 years old or older, being diagnosed of any kind of EPILEPSY (criteria ILAE) and with diagnosis being confirmed by a Neurologist over the last 6 months and with write informed consent.

Exclusion Criteria:

* Patients with epilepsy diagnosis confirmed by a Neurologist over the last 6 months before the study or with incapacity to fulfill the requirements of the study.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients being diagnosed of any kind of EPILEPSY (criteria ILAE 2005) and with diagnosis being confirmed by a Neurologist over the last 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2008-02; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (1):
- UCB Pharma, Smyrna, Georgia, United States